CLINICAL TRIAL: NCT04288648
Title: Pelvic Floor Contraction in Different Positions Among Women With and Without Stress Urinary Incontinence
Status: Completed | Type: Observational
Sponsor: University of Haifa (Other)
Responsible Party: Principal Investigator, Gali Dar, principal investigator, University of Haifa
Other Study IDs: HU 26/2020
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Urinary Stress Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SUI group: Examination will include an abdominal ultrasound assessment of pelvic floor muscle in supine, sitting, standing and squatting. The Height of the bladder base will be measured during rest period and maximal contraction.
  Interventions: Diagnostic Test: ultrasound examination
- control group: Examination will include an abdominal ultrasound assessment of pelvic floor muscle in supine, sitting, standing and squatting. The Height of the bladder base will be measured during rest period and maximal contraction.
  Interventions: Diagnostic Test: ultrasound examination

INTERVENTIONS:
Diagnostic Test: ultrasound examination — ultrasound examination of pelvic floor muscle will be conducted. In addition questionnaires regarding demographic characteristics and SUI will be performed.
  Other Names: transabdominal ultrasound assessment

SUMMARY:
Examination of pelvic floor contraction in different positions among women with and without stress urinary incontinence (SUI) will be conducted via diagnostic ultrasound. This will enable clinicians and researchers to establish an appropriate protocol for pelvic floor muscle examination and treatment.

DETAILED DESCRIPTION:
The main goal of this study is to compare the ability of the pelvic floor muscles to contract in different positions among women suffering from SUI to healthy women. Secondary objectives: is to compare subjective reports of the difficulty to contract the pelvic floor muscles between the two groups, and to examine the connection between the severity of urinary leakage and the ability to contract pelvic floor muscles.

The study will include 50 female participants in the ages of 18-45. Research group will include 25 participants suffering from SUI in accordance with the International Consultation on Incontinence Questionnaire Short Form (ICIQ-SF) and 25 healthy participants (grade 0 on the ICIQ-SF questionnaire).

The examination will be performed with an abdominal ultrasound device in supine, sitting, standing and squatting. The Height of the bladder base will be measured during rest period and maximal contraction. The extent and direction of bladder base movement would indicate the quality of pelvic floor performance. Next, the length of contraction time will be measured. The participant would hold the maximal contraction as long as possible in order to examine muscular endurance. Rest will be given between tests. After finishing the tests in all four postures, the participants will be questioned about the degree of difficulty contracting the pelvic floor.

Significance of the study: The importance of the research is about granting the clinicians and researchers additional tools in order to help establishing a protocol for pelvic floor muscle activity examination and treatment.

ELIGIBILITY:
Inclusion Criteria (general):

* willing to participate in the study
* being able to squat for over 10 seconds.
* inclusion for study group - participants suffering from SUI that received a grade>0 in sections 3+4 (how frequent does urinary leakage appear, the amount of urine leakage and does the participant use pads for leakage absorption) and a grade>0 in section 5 (how much does SUI interrupt the participant's daily life) in the International Consultation on Incontinence Questionnaire Short Form (ICIQ-SF).
* Inclusion for control group - healthy participants (grade 0 in the ICIQ- SF questionnaire).

Exclusion Criteria:

* Other types of urinary leakage
* receiving pelvic floor treatments in the past or present
* active urinary or vaginal infections
* neurological diseases
* urologic, gynecologic or abdominal surgery
* pelvic organ prolapse
* pregnancy
* chronic cough
* constipation
* unbalanced diabetes and the use of medication that affects urination

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — women only
Study Population: Women, between ages 18-45 with and without USI.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2020-05-17 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
direction of urinary bladder displacement during contraction | baseline
  upward or downward displacement of urinary bladder will be measured via diagnostic ultrasound

SECONDARY OUTCOMES:
urinary bladder displacement in millimeters | baseline
  bladder displacement will be measured via diagnostic ultrasound using the on screen caliper tool
pelvic floor muscles endurance of contraction in seconds | baseline
  time of muscle contraction will be measured during the last contraction
questioned about the degree of difficulty contracting the pelvic floor. | baseline
  Each participant will grade on a scale of 1-10 (10 most difficult) the subjective difficulty of contraction in each position

CONTACTS AND LOCATIONS:
Overall Officials: Gali Dar, PhD, Principal Investigator — Gali Dar, Department of Physical Therapy, University of Haifa
Locations (1):
- Haifa University, Department of PHysical Therapy, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Yes
following study completion, a paper will be submitted to international professional journal
Supporting Information: Study Protocol, SAP
Time Frame: 6 months following end of study

REFERENCES:
- [Result] Sapsford RR, Richardson CA, Stanton WR. Sitting posture affects pelvic floor muscle activity in parous women: an observational study. Aust J Physiother. 2006;52(3):219-22. doi: 10.1016/s0004-9514(06)70031-9. PMID 16942457